CLINICAL TRIAL: NCT02257697
Title: A Multi-center, Randomized, Controlled, Open-label Clinical Study to Evaluate the Efficacy and Safety of Mizoribine in Comparison With Cyclophosphamide in the Treatment of Refractory Nephrotic Syndrome
Brief Title: A Study to Evaluate the Efficacy and Safety of Mizoribine in the Treatment of Refractory Nephrotic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asahi Kasei Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE-69-C-Ne-302
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — mizoribine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mizoribine (MZR) (Experimental): Oral administration, daily dose of 150mg (50mg/tablet, t.i.d) All study subjects will receive standard steroid therapies during the study.
  Interventions: Drug: Mizoribine (MZR)
- Cyclophosphamide (CTX) (Active Comparator): Intravenous injection with between 0.5 to 1.0 g/m2 body surface area each time (the maximum dose is 1.0 g/day each time).
  All study subjects will receive standard steroid therapies during the study.
  Interventions: Drug: Cyclophosphamide (CTX)

INTERVENTIONS:
Drug: Mizoribine (MZR)
  Other Names: HE-69
  Arms: Mizoribine (MZR)
Drug: Cyclophosphamide (CTX)
  Arms: Cyclophosphamide (CTX)

SUMMARY:
To demonstrate that the treatment effect in refractory nephrotic syndrome of MZR is non-inferior to that of standard therapy CTX through analyzing overall remission rate after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have medical history with clear documentation of diagnosis of nephrotic syndrome
* Patient who received renal biopsy within 1 year prior to screening and confirmed the pathologic classification: Minimal Change Disease (MCD), IgA nephropathy, Mesangioproliferative Glomerulonephritis (MsPGN), Membranous Nephropathy (MN), Focal Segmental Glomerulosclerosis (FSGS)
* Patient with the above different pathologic classification who received adequate hormone therapy more than 8 weeks (including FSGS more than 12 weeks)prior to screening and have 24hr-urine protein≥2.0g/day at screening Adequate hormone dose is defined as prednisone (prednisolone) equivalent dose of 0.8 to 1.0 mg/kg/day (inclusive)
* Male or female patient between 18 and 70 years (inclusive) at informed consent obtained date
* Patient with body weight between 40kg and 80kg (inclusive) at screening
* Patients who sign the informed consent form

Exclusion Criteria:

* Other primary nephrotic syndrome, e.g. membrano-proliferative glomerulonephritis (MPGN)
* Secondary nephrotic syndrome (e.g. diabetic nephropathy, anaphylactic purpura nephritis, lupus nephritis, type B hepatitis-related nephritis, renal amyloidosis)
* Patient who had history of allergy to any investigational product (MZR, CTX) or hormone
* Patient who had received accumulated dosage of CTX >3g within one year prior to screening
* Patient who had received immunosuppressant or Chinese traditional medicine with immunosuppressive effect within 30 days prior to screening
* Patient who received other investigational drugs within 30 days prior to screening
* Patient who have received plasma exchange therapy or immunoadsorption therapy within 30 days prior to screening
* Patient who require pentostatin or live vaccine (not including flu vaccine)
* Patient who is undergoing renal replacement therapy
* Patient who received kidney transplantation
* Patient with malignancy
* Patient with severe hypertension (SBP > 160mmHg or DBP > 100mmHg) which has not been effectively controlled
* Patient with white blood cell count <3×109/L /L(=3.0 GI/L)
* Patient with SCr > 176.8μmol/L
* Patient who has a value that is > 3 times of the upper limit of normal range for AST or ALT
* Patient with hepatitis B, hepatitis C or HIV infection
* Patient with other serious infections
* Patient who is unsuitable for participating in this study in the opinion of investigators ( e.g. uncontrolled diabetes, central nervous system lupus , lupus encephalopathy, active psychosis,osteonecrosis of the femoral head, fulminant hepatitis, peptic ulcer, etc.)
* Female patient who is pregnant, currently breast feeding or willing to become pregnant
* Patient with any other diseases that would affect the evaluation of efficacy or safety

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2014-11; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Total Remission rate | 52 weeks

SECONDARY OUTCOMES:
Complete Remission rate | 52 weeks
Partial Remission rate | 52 weeks
Changes of Overall Remission rate | 8 weeks, 20 weeks, 32 weeks, 44 weeks and 52 weeks
Changes of Complete Remission rate | 8 weeks, 20 weeks, 32 weeks, 44 weeks and 52 weeks
Changes of Partial Remission rate | 8 weeks, 20 weeks, 32 weeks, 44 weeks and 52 weeks
Treatment failure rate | 52 weeks
Changes and percentage change of 24 hours urine protein and serum albumin from the baseline | 8 weeks, 20 weeks, 32 weeks, 44 weeks and 52 weeks
Changes of and percentage change of SCr, eGFR and BUN from the baseline | 8 weeks, 20 weeks, 32 weeks, 44 weeks and 52 weeks
Progression to End-Stage Renal Disease or Doubling of SCr through the study | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Asahi Kasei Pharma Corporation, Study Chair — Asahi Kasei Pharma Corporation
Locations (28):
- China (28):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The Third Affiliated Hospital of the Third Military Medical University (Daping Hospital), Chongqing, Chongqing Municipality
  - Fuzhou General Hospital of Nanjing Military Region, Fuzhou, Fujian
  - The first Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The General Hospital of Shenyang Military Region, Shenyang, Liaoning
  - Shandong Provincial Hospital, Jinan, Shandong
  - The General Hospital of Jinan Military Region, Jinan, Shandong
  - The Affilited Hospital of Qingdao University, Qingdao, Shandong
  - Renji Hospital Shanghai Jiaotong University School of Medical, Shanghai, Shanghai Municipality
  - Xinhua Hospital Shanghai Jiaotong University School of Medical, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - The Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xian, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Kuming General Hospital of Chengdu Military Region, Kunming, Yunnan
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Dong Z, Zhou J, Xu Z, Ni Z, He Y, Lin H, Jiang G, Sun X, Zhang L, Chen X. Efficacy and Safety of Mizoribine for the Treatment of Refractory Nephrotic Syndrome: Protocol for a Multicenter, Controlled, Open-label, Randomized Controlled Trial. JMIR Res Protoc. 2023 Jun 16;12:e46101. doi: 10.2196/46101. PMID 36990111